CLINICAL TRIAL: NCT00359346
Title: Plasma Exchange for Autoimmune Autonomic Failure
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060209; 06-N-0209
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-16

CONDITIONS: Plasma Exchange; Autonomic Failure
Keywords: Plasmapheresis; Auto-antibodies; Autonomic Nervous System; Dysautonomia; Sympathetic Nervous System; Autonomic Failure
MeSH Terms: conditions — Pure Autonomic Failure; Autonomic Nervous System Diseases

SUMMARY:
This study will explore whether an antibody is influencing the autonomic nervous system, and if its removal will eliminate signs and symptoms of failure in that system. The autonomic nervous system is responsible for many automatic changes involved in everyday activities, such as standing up, digesting food, and exercising in the heat. Antibodies fight germs but sometimes cause health problems. Removal of the antibody is done through a procedure called a plasma exchange.

Patients with primary chronic autonomic failure and a circulating antibody to what is called the neuronal nicotinic receptor may be eligible for this study. To be eligible, patients will have participated in an earlier study, protocol number 03-N-0004. Patients will undergo tests and procedures that include an electrocardiogram, and blood collection for hepatitis, HIV, and pregnancy. Blood will be tested for a complete blood count, clotting factors, and chemistries. There will also be tests for liver function, kidney function, cortisol, and thyroid. Participants will be tested for signs and symptoms of autonomic failure, and will be asked to complete questionnaires about various symptoms before the plasma exchange, 1 or 2 weeks afterward, and then monthly or bimonthly for up to 1 year. Patients will undergo a series of other tests. In one test, a patient is upright and blows against a resistance (Valsalva maneuver). The quantitative sudomotor axon reflex test (QSART) uses iontophoresis, involving application of acetylcholine, a chemical messenger, and a small amount of electricity. QSART examines the regulation of sweating, a particular aspect of the autonomic nervous system. There will be a test using edrophonium, given intravenously (IV), to evaluate that drug's effects on the heart, skin, glands, gastrointestinal activity, bladder tone, and salivation. A glucagon test, also by IV, will show patients' ability to release the hormone adrenaline.

The plasma exchange will be performed by use of an automated cell separator. Patients' blood will be removed continuously through a needle in the arm. Blood cells will be separated from the plasma by a spinning process and continuously returned to circulation through a needle in the patients' opposite arm. Blood cells that are returned will be mixed with albumin, a sterile replacement solution. A blood thinner, citrate, will be given, to prevent clotting of blood. This whole procedure will take about 2 hours. Patients will typically undergo five exchange procedures in about 10 days while they are inpatients at the NIH Clinical Center. The amount of plasma removed in a single session and the number of sessions will be set by the NIH Blood Bank. It is expected that patients' autonomic failure will improve after several days of starting the plasma exchange. Testing for symptoms of autonomic failure and autonomic function testing will occur about 1 month after the plasma exchange and monthly or bimonthly for up to 1 year. For each visit of testing, patients will be inpatients for about 2 days. If autonomic failure recurs, patients may have a second plasma exchange, with the same follow-up tests, for about 1 year.

DETAILED DESCRIPTION:
Background: Until recently, it was thought that primary chronic autonomic failure occurring without central neurodegeneration (pure autonomic failure, PAF) reflected diffuse loss of catecholamine-producing cells (sympathetic noradrenergic nerves and adrenomedullary chromaffin cells) outside the brain. Rarely, however, PAF patients have clinical laboratory findings suggesting decreased post-ganglionic nerve traffic in intact autonomic nerves, rather than denervation. To date, all of four such patients have also had a high titer of a circulating antibody to the nicotinic receptor mediating ganglionic neurotransmission. In one case, studied by another group, plasma exchange reversed signs and symptoms of autonomic failure, consistent with the antibody being pathogenic.

Purpose: In this Protocol, we will carry out plasma exchange in patients we identify as having PAF, intact cardiac noradrenergic innervation, and a circulating antibody to the neuronal nicotinic receptor, to determine whether antibody pathogenicity is a consistent finding in this condition. We will assess the extent of relationship between symptoms, signs, and clinical laboratory indices of autonomic function with the titer of the antibody and obtain abundant plasma for antibody characterization and target protein identification.

Methods: Autonomic function testing will be done before plasma exchange, 1-2 weeks after plasma exchange, and monthly or bi-monthly thereafter for up to one year. Plasma exchange may be repeated once, when symptoms of autonomic failure return as the antibody level builds up, to verify in individual patients whether repetition of plasma exchange produces reproducible amelioration of clinical and laboratory measures of autonomic failure.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects have primary chronic autonomic failure, intact cardiac sympathetic innervation, and a circulating antibody to the nicotinic cholinergic receptor mediating ganglionic neurotransmission. This triad will be identified based on results of participation in NIH Clinical Protocol 03-N-0004.

EXCLUSION CRITERIA:

Subjects are excluded if they do not meet all three of the above Inclusion Criteria.

Venous Access Candidate subjects are excluded if there is inadequate peripheral venous access, identified during participation in NIH Clinical Protocol 03-N-0004.

Abnormal Clinical Pathology Test Results Candidate subjects are excluded based on abnormal Clinical Pathology results identified during participation in NIH Clinical Protocol 03-N-0004 (platelet count less than 100,000 per microliter, HIV-1 or 2 or chronic hepatitis B or C infection, or pregnancy).

Medical Risk Candidate subjects are excluded for safety reasons if, in the opinion of the Associate Investigator of the NIH Department of Transfusion Medicine (DTM), therapeutic plasma exchange would pose an excessive risk of complications (e.g., stroke, hemorrhage, infection) outweighing the potential scientific and clinical benefit. In female patients with child-bearing potential, a blood test for pregnancy is done prior to testing on each visit. The finding of a positive test for pregnancy excludes the patient from further participation.

Patients with autonomic failure have an increased risk of hypotension in response to manipulations that decrease venous return to the heart, such as plasma exchanges. Patients with autonomic failure typically also have high blood pressure when they are lying down. We expect that at the beginning of plasma exchanges, the blood pressure will be relatively high, and the plasma exchanges may be started with the patient in a sitting position. The Principal Investigator or one of the other Associate Investigators of the Clinical Neurocardiology Section will monitor the blood pressure frequently or continuously during the plasma exchanges. Patients with autonomic failure often tolerate remarkably low blood pressure. A systolic blood pressure of 90 mm Hg will be the threshold for intervening. The first intervention will be to place the patient in a supine position. Second, we would administer saline and albumin and slow down the rate of or stop the plasma exchange. Drugs to control blood pressure will also be on hand for immediate emergency use if needed. If we think that we cannot prevent low blood pressure and fainting during future plasma exchanges, then we would exclude the patient from further plasma exchanges under this Protocol. If uncontrollable hypotension occurs in a second patient, then the Protocol will be terminated.

Patients are tested for hepatitis and for HIV before undergoing plasma exchange. Blood from people with hepatitis or HIV can contaminate the Blood Bank equipment. If a subject has hepatitis or HIV, the subject will be excluded from further participation in the study. The Consent Form includes standard consent language about HIV testing.

Age - The Protocol is restricted to subjects at least 18 years old.

Medications - Medications likely to interfere with the scientific results will be discontinued on an inpatient basis.

Termination of Participation - A subject may refuse certain tests or procedures, or may terminate participation early, without loss of benefits to which the subject was previously entitled. The Investigators may also exclude a subject from further participation, such as in the event of known or suspect falsification of medical history information or refusal to undergo planned tests or procedures, without loss of benefits to which the subject was previously entitled.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3
Dates: Start 2006-07-14; Study Completion 2009-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ziegler MG, Lake CR, Kopin IJ. The sympathetic-nervous-system defect in primary orthostatic hypotension. N Engl J Med. 1977 Feb 10;296(6):293-7. doi: 10.1056/NEJM197702102960601. PMID 831126
- [Background] Goldstein DS, Holmes C, Dendi R, Li ST, Brentzel S, Vernino S. Pandysautonomia associated with impaired ganglionic neurotransmission and circulating antibody to the neuronal nicotinic receptor. Clin Auton Res. 2002 Aug;12(4):281-5. doi: 10.1007/s10286-002-0020-3. PMID 12357282
- [Background] Schroeder C, Vernino S, Birkenfeld AL, Tank J, Heusser K, Lipp A, Benter T, Lindschau C, Kettritz R, Luft FC, Jordan J. Plasma exchange for primary autoimmune autonomic failure. N Engl J Med. 2005 Oct 13;353(15):1585-90. doi: 10.1056/NEJMoa051719. PMID 16221781